CLINICAL TRIAL: NCT01206231
Title: An Epidemiological Study Aimed to Record Standard Daily Practice in Managing Patients With Hypercholesterolemia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRS-DUM-2010/1
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypercholesterolemia
Keywords: Standard daily practice in managing patients with hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hypercholesterolemia

SUMMARY:
This study is aimed to collect the following Serbia-specific epidemiology data on hypercholesterolemia: patents characteristics, patients' management/treatment and physicians' standard practice. In addition, the aim is to determine the proportion of patients on lipid-lowering pharmacological treatment who have reached the LDL-C and HDL-C treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypercholesterolemia currently receiving a lipid lowering agent

Exclusion Criteria:

* Pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality care clinics
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the NCEP ATP III / updated 2004 NCEP ATP III guidelines | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients on lipid-lowering pharmacological treatment reaching the non HDL-C goals according to the NCEP ATP III / updated 2004 NCEP ATP III guidelines; | 24 weeks
Physicians' standard practice in managing patients with hypercholesterolemia (by using physicians' questionnaire); | 24 weeks
Local epidemiological date on patients with hypercholesterolemia (Demographic Data; Hypercholesterolemia management data: treatment, treatment changes) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr Miodrag Ostojic, Principal Investigator — Division of Cardiology-Clinical Centre of Serbia-Belgrade
Locations (10):
- Serbia (10):
  - Research Site, Belgrade
  - Research Site, Čačak
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Niška Banja
  - Research Site, Pančevo
  - Research Site, Požarevac
  - Research Site, Sombor
  - Research Site, Užice